CLINICAL TRIAL: NCT05494866
Title: IntenSify: an Open-label Phase I Trial of the CYP3A Inhibitor Cobicistat and the Cytostatics Gemcitabine and Nab-Paclitaxel in Patients with Advanced Stage or Metastatic Pancreatic Ductal Adenocarcinoma to Evaluate the Combination's Pharmacokinetics, Safety and Efficacy
Brief Title: A Trial of Cobicistat and Gemcitabine and Nab-Paclitaxel in Patients with Advanced Stage or Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: IntenSify
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of efficacy paired with high toxicity
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NH21; 2019-001439-29 (EudraCT Number)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: CYP3A Inhibitor; Advanced Stage or Metastatic Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreatic Neoplasm
Keywords: CYP3A Inhibitor; Pancreatic Ductal Adenocarcinoma; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Cobicistat; Anti-HIV Agents; Anti-Retroviral Agents; Antiviral Agents; Anti-Infective Agents; Cytochrome P-450 CYP3A Inhibitors; Cytochrome P-450 Enzyme Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms | interventions — Cobicistat; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): CYP3A Inhibitor Cobicistat and the cytostatics Gemcitabine and nab-Paclitaxel
  Interventions: Drug: Cobicistat Oral Tablet; Drug: Gemcitabin; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Cobicistat Oral Tablet — Cobicistat Oral Tablet
Drug: Gemcitabin — Gemcitabin
Drug: Nab paclitaxel — nab-Paclitaxel

SUMMARY:
To explore the possibility to overcome CYP3A-mediated resistance to anticancer drugs in pancreatic cancer, we will investigate the pharmacokinetics, safety, tolerability, and efficacy of nanoparticle albumin-bound paclitaxel (nab-paclitaxel) in combination with gemcitabine and the CYP3A inhibitor cobicistat in a phase I proof-of-concept trial to determine the safety profile, the recommended dose of nab-paclitaxel in combination with gemcitabine and cobicistat, and to determine whether there is an early efficacy signal warranting a larger scale trial.

The present trial is an open-label trial consisting of a dose-escalation part and an expansion part. The dose escalation part is designed to determine the safety, tolerability, and pharmacokinetics of nab-paclitaxel in combination with gemcitabine and cobicistat and will guide the dosing in the expansion part of the trial.

The trial enrolls patients with unresectable locally advanced or metastatic pancreatic adenocarcinoma and adequate performance score (ECOG PS 0-2) who would usually receive gemcitabine and nab-paclitaxel according to standard of care.

Primary endpoint for the phase I trial is the safety of the combination. Overall survival (OS), disease control rate (DCR), overall response rate (ORR), duration of response (DoR) and progression free survival (PFS) are secondary efficacy endpoints. Further secondary endpoints are tolerability, pharmacokinetics, pharmacodynamics, and pharmacogenomics.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years
2. Histologically or cytologically confirmed ductal adenocarcinoma of the pancreas.
3. Metastatic disease. Advanced stage locally advanced, unresectable (patients that are resectable but refuse the operation are not eligible) may be eligible after discussion with the medical representative of the sponsor
4. Eligible for therapy with gemcitabine / nab-paclitaxel according to standard of care / local therapeutic standard (in any palliative therapy line)
5. Performance score ECOG 0-2
6. Adequate organ function defined as:

   1. Adequate hematologic function (WBC ≥3000/µL, absolute neutrophil count ≥1500/µL, platelets ≥100.000/µL, hemoglobin ≥8 g/dL)
   2. Adequate renal function (estimated glomerular filtration rate ≥30 mL/min)
   3. Adequate liver function (serum bilirubin ≤1.5 x ULN, AST/ALT ≤2.5 x ULN, or 5 x ULN if hepatic metastases are present)
   4. Prothrombintime (PT) <1.1 ULN, partial thromboplastin time <1.1 ULN, INR <1.1 ULN.
7. Use of reliable contraception with a Pearl Index <1% (i.e. two independent effective contraceptive methods) during the trial and for two weeks after the last administration of trial medication in men or women of child bearing potential (WOCBP).
8. Measurable disease according to RECIST 1.1 criteria.
9. Patient willing to undergo tumor biopsy. This requires a tumor lesion accessible for a biopsy. In patients without an accessible tumor lesion the patient may be enrolled and tumor biopsy waived after discussion with the sponsor's medical representative.
10. Available CT scan of thorax and abdomen not older than 30 days before start of treatment (day 1 of cycle 1). Patients that cannot have a CT scan because of medical reasons (e.g. allergy to contrast dye) may be eligible after MRIs as per standard of care to stage the patient and after documented consultation with the sponsor.
11. Ability to understand character, consequences and requirements of the clinical trial and to comply with the study protocol and dosing regimen.

Exclusion Criteria

1. Presence of brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
2. Testing positive against human immunodeficiency virus (HIV) or history thereof
3. Active hepatitis C virus (HCV) infection (patients with status post-infection after eradication through antiviral therapy are eligible)
4. Uncontrolled hepatitis B virus (HBV) infection (<3 months of treatment with a nucleotide analogue and/or >100 HBV-DNA particles)
5. Pre-existing, clinically significant peripheral neuropathy, defined as CTCAE grade 2 or higher neurosensory or neuromotor toxicity, regardless of etiology
6. History of malignancy other than pancreatic cancer in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
7. Present treatment with phenprocoumon, warfarin or another coumadine-based anticoagulant.
8. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
9. Major surgery, other than for diagnostic purposes ((done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
10. History of allergy or hypersensitivity to any of the study drugs or any of their excipients.
11. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise patient's safety or study data integrity.
12. Participation in any other interventional clinical protocol or investigational trial.
13. Unwillingness or inability to comply with study procedures.
14. Therapy with a narrow therapeutic index drug that is substrate of CYP3A, CYP2D6, or CYP2C9 whose dose cannot be appropriately adjusted.
15. Therapy with any medications or substances that are inhibitors or inducers of CYP450 3A enzyme(s) or therapy with medication that is contraindicated when taking Tybost
16. Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
occurrence of DLTs | Day 1 to day 28
  occurrence of DLTs within treatment cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Hohmann, PD Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hohmann N, Sprick MR, Pohl M, Ahmed A, Burhenne J, Kirchner M, Le Cornet L, Kratzmann M, Hajda J, Stenzinger A, Steindorf K, Delorme S, Schlemmer HP, Riethdorf S, van Schaik R, Pantel K, Siveke J, Seufferlein T, Jager D, Haefeli WE, Trumpp A, Springfeld C. Protocol of the IntenSify-Trial: An open-label phase I trial of the CYP3A inhibitor cobicistat and the cytostatics gemcitabine and nab-paclitaxel in patients with advanced stage or metastatic pancreatic ductal adenocarcinoma to evaluate the combination's pharmacokinetics, safety, and efficacy. Clin Transl Sci. 2023 Dec;16(12):2483-2493. doi: 10.1111/cts.13661. Epub 2023 Nov 3. PMID 37920921